CLINICAL TRIAL: NCT03753594
Title: Changes of Regional Tissue Oxygenation Saturation After Successful Femoral Nerve Block With Ropivacaine at Different Concentrations
Brief Title: Changes of Regional Tissue Oxygenation Saturation After Successful Femoral Nerve Block
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xi Wu, Principal Investigator, Department of Anesthesiology, Union Hospital of Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XH20181118
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Anesthesia, Local
Keywords: Peripheral nerve block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- H group: Patients scheduled for elective knee arthroscopy with peripheral nerve block will receive ultrasound-guided femoral nerve block with 0.5% ropivacaine. Regional tissue oxygenation saturation of the nerve innervation area and pinprick sensory tests at 5 min were assessed before the block and at 5-min intervals till 30 min after the block.
  Interventions: Device: tissue oxygenation saturation
- L group: Patients scheduled for elective knee arthroscopy with peripheral nerve block will receive ultrasound-guided femoral nerve block with 0.25% ropivacaine. Regional tissue oxygenation saturation of the nerve innervation area and pinprick sensory tests were assessed at 5 min before the block and at 5-min intervals till 30 min after the block.
  Interventions: Device: tissue oxygenation saturation

INTERVENTIONS:
Device: tissue oxygenation saturation — tissue oxygenation saturation

SUMMARY:
Regional tissue oxygenation saturation has been shown to increase in innervated regions after sympathetic block. The aim of this prospective observational study was to evaluate the changes of regional tissue oxygenation saturation by near-infrared spectroscopy after successful femoral nerve block with ropivacaine and determine whether the changes of regional tissue oxygenation saturation can be affected by the concentration of ropivacaine.

DETAILED DESCRIPTION:
Successful peripheral nerve blocks induce sympathetic blockade, which increases local blood flow by vasodilation. The relationship between successful femoral nerve block and the variation of regional tissue oxygenation saturation was unclear.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* American Society of Anesthesiologists physical statusⅠ-Ⅱ
* Undergo elective elective knee arthroscopy with peripheral nerve block

Exclusion Criteria:

* Refusal to participate in the study
* BMI>35
* Any contraindications to peripheral nerve block such as coagulation abnormalities, •Allergy to local anaesthetics, peripheral neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred adult patients scheduled for elective knee arthroscopy with peripheral nerve block
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Regional tissue oxygenation saturation after successful femoral nerve block | at 5-minute intervals till 30 minutes after regional block
  rSO2

SECONDARY OUTCOMES:
Pinprick sensory scores | 5 minute before regional block and at 5-minute intervals till 30 minutes after regional block
  A 3-level scale was used to grade the intensity of sensory block using pinprick stimulation: 0=normal sensation; 1=analgesia; 2=anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Chen, Doctor, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Wuhan, Hubei, China